CLINICAL TRIAL: NCT06464250
Title: The Effect of Bundle Approach on Foot Care Behaviors and Wound Healing in Patients Applying to Diabetic Wound Outpatient Clinic
Brief Title: The Effect of Bundle Approach on Foot Care Behaviors and Diabetic Wound Healing in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Cıgdem Yavuz Batmaz, Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DYCYBHBK01
Record Dates: First submitted 2024-05-21; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Wound; Diabetic Foot Ulcer; Ulcer
Keywords: Diabetic Foot; Diabetic Foot Ulcer; Wound; Ulcer; Bundle; Care Package Approach
MeSH Terms: conditions — Wounds and Injuries; Diabetic Foot; Ulcer

STUDY DESIGN:
Intervention Model Description: In the study, there are two parallel groups as control and intervention groups.
Who Masked: Participant
Masking Description: In the study, participant blinding was performed by ensuring that the participants did not know which group they were in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bundle care group (Experimental): Before the intervention, both the Control and Intervention groups underwent face-to-face interviews and completed forms such as the 'Patient Identification Form,' 'Nottingham Functional Foot Care Diagnosis Form,' and 'Diabetic Foot Evaluation Form.' Subsequently, both groups received one-on-one training covering various aspects related to diabetic foot. This training, conducted by the researcher, involved interactive question-answer sessions and practical demonstrations of foot care techniques.
  Following the training, the Intervention group received a care package comprising foot examination, guidance on correct foot care practices, and a request for regular blood glucose monitoring. These patients were then monitored at the 1st, 2nd, and 3rd months.
  Interventions: Other: Bundla care group
- Control Group (No Intervention): For the Control group, after receiving education and brochures, the 'Nottingham Functional Foot Care Diagnostic Form' and 'Diabetic Foot Evaluation Form' were completed at the 1st, 2nd, and 3rd months. Similar to the Intervention group, new wound formation, wound classification, and healing status of existing ulcers were monitored for this group as well.

INTERVENTIONS:
Other: Bundla care group — A care package consisting of foot examination, correct foot care behaviours, and regular blood glucose monitoring was used.
  Arms: Bundle care group

SUMMARY:
This study was planned to standardize foot care behaviors with a patient-participated care package approach, to ensure healing of existing wounds, and to evaluate the effect on foot care behaviors to prevent the development of new diabetic foot ulcers. The sample of the study consisted of a total of 97 patients, 49 patients in the care package group and 48 patients in the control group.

Hypotheses of the Study H1. The foot care behaviors of patients who receive a patient-participatory care package approach to diabetic foot ulcer prevention will be higher than those of patients who do not receive a care package.

H2. Patient-involved care package approach prevents the development of new diabetic foot ulcers.

H3. Patient-involved care package approach provides healing of existing diabetic ulcers.

DETAILED DESCRIPTION:
The research was planned as a randomized controlled experimental study to standardize foot care behaviors with a care package approach consisting of evidence-based practices for patients with diabetic ulcers who applied to Başakşehir Çam and Sakura City Hospital diabetic wound outpatient clinic in Istanbul, to ensure healing of existing wounds, to prevent new diabetic foot ulcers, and to evaluate the effect on foot care behaviors. The average number of patients with diabetic foot ulcers 1-2 and 3 according to the Wagner classification is 300 people. According to the Power analysis (G*Power 3.1.9.7), it was aimed to reach at least 95 people in total with an effect size of 0.458, 5% margin of error and 95% power.Data were collected by the researcher through face-to-face interviews with the patient. "Patient Identification Form", "Nottingham Functional Foot Care Diagnosis Form (NAFF)", "Diabetic Foot Evaluation and Follow-up Form" were used. The patient identification form consists of 17 questions as a result of literature review. The Nottingham Assessment of Functional Footcare (NAFF) was developed by Lincon et al. in 2007 and focuses on foot care behaviors. "Diabetic foot assessment and follow-up form" was created by the researcher and the depth, length and width of the wound were measured to observe whether new wounds were formed and the healing status of the wound. Spearman Correlation Test was used to analyze the measured data with each other. P-values below 0.05 were considered as statistically significant results.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* No reading and comprehension problems,
* No psychiatric disorders,
* Wounds with Wagner 1-2 and 3 according to the Wagner classification (
* Individuals who agreed to participate in the study.

Exclusion Criteria:

* Under 18,
* Wounds other than diabetic ulcers,
* Wounds with Wagner 4 and Wagner 5 according to the Wagner classification (this wound class includes ischemic wounds),
* Below/above knee amputation in the limb other than the at-risk/injured foot,
* Psychiatric problems,
* Refuses to work or wants to leave during the work,
* Individuals with reading and comprehension problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
individual benefit | at the end of three months
  It is useful for individuals with diabetic foot wounds to gain positive behaviors and reduce the development of complications.Through the Nottingham Assessment of Functional Footcare (NAFF), it is assessed that the individual gains positive foot care behaviors. The existing wound of the individual who gains positive foot care behaviors improves, new wound formation is prevented, and diabetes is controlled. The Nottingham Assessment of Functional Footcare (NAFF) is based on individuals' responses on four Likert-type scales of foot care behavior, with each item scored from zero to three. A high score indicates positive foot care behavior.
social benefit | at the end of three months
  The care package approach aims to reduce the development of diabetic foot ulcers in the community.The diabetic foot assessment and follow-up form was used to measure the depth, length and width of the wound to observe whether new wounds were formed and the healing status of the wound. The commonly used Wagner classification, which facilitates wound classification by grading the wound from 0 to 5, was used.With the care package approach, the individual knows the factors that may cause new wounds as a result of the positive behaviors he/she gains and prevents the formation of new wounds by behaving accordingly.
scientific utility | at the end of three months
  The results of the literature review will contribute to further studies with individuals with diabetic foot ulcers and to the evaluation of the effectiveness of the care bundle approach. The care package has been studied in different fields but has been limited to individuals with diabetic foot. After the literature review and expert opinion, the effect of the care package on the foot care behaviors of patients with diabetes in the "Patient-participated diabetic foot ulcer preventive care package" will be evaluated on new wound formation and wound healing. Face-to-face data will be collected. "Nottingham Assessment of Functional Footcare" scale will be used for foot care behaviors and "Wagner classification" will be used for wound assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Yavuz Batmaz, Principal Investigator — Marmara University
Locations (1):
- Başakşehir Çam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)